CLINICAL TRIAL: NCT04184011
Title: A Prospective Registry Study to Evaluate the Long-Term Efficacy and Safety of Superficial Radiation Therapy (SRT) for the Treatment of Recurrent Keloid Scars
Brief Title: Superficial Radiation Therapy (SRT) for the Treatment of Recurrent Keloid Scars
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sensus Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: SRTS-SRT-003
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Keloid Scar
Keywords: Superficial Radiation Therapy
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SRT for keloid scars: Individuals who are voluntarily scheduled to be treated at one of the participating study sites with SRT (SRT-100™, SRT-Vision™ or SRT-100+™) for the treatment of one or more recurrent keloids.
  Interventions: Device: SRT-100™

INTERVENTIONS:
Device: SRT-100™ — SRT delivers a precise, calibrated dose of radiotherapy following surgical excision for large and more difficult-to-treat keloids that cannot otherwise be treated by or have failed more conservative measures.

SUMMARY:
Keloid formation in response to skin trauma inflicts about 18 million individuals. A key impediment in successful treatment of keloids is that the predominant treatments, particularly surgical excision and shaving, tend to initiate the regrowth of the keloid at the excision site, and therefore, recurrence rates are high. There is much evidence to demonstrate that following surgical excision procedures with a course of radiation therapy can significantly reduce recurrence rates to as little as 10% or below. This prospective study is to evaluate this claim.

DETAILED DESCRIPTION:
A keloid is an unsightly non-malignant tumor comprised of an abnormal proliferation of scar tissue that forms at the site of cutaneous injury (e.g. skin trauma such as cuts, abrasions and puncture wounds, burns or surgical incisions). It appears as a raised scar and does not regress and grows beyond the original margins of the scar. Keloids most commonly develop on the earlobes, neck, shoulders, chest, back, upper arms and cheeks. Keloids tends to grow slowly and continue to spread for weeks, months or even years. As a keloid grows, it may cause significant itching, pain, and tenderness upon touch, reduced mobility and emotional distress.

About 18 million people worldwide are genetically prone to form keloids in response to skin trauma, with equal gender distribution and greater susceptibility for darker-skinned individuals and those aged 10 to 30 years.

The greatest obstacle in treating keloids with many available surgical and non-surgical methods is that new keloids typically recur at the site of excision due to the treatment itself. For example, the recurrence rate using surgical excision alone is 45 to 100 percent.

Surgical excision followed by radiotherapy is a helpful treatment option for large and more difficult-to-treat keloids that cannot otherwise be treated by, or have failed, more conservative measures. It is thought that because keloid fibroblasts are sensitive to x-ray irradiation, it may prevent the recurrence of keloids by controlling fibroblast proliferation, arresting the cell cycle, and inducing premature cellular senescence. When surgical keloid excision is followed by Radiation Therapy, recurrence drops dramatically to 10% or below.

The SRT-100™ is a United States Food and Drug Administration (U.S. FDA) approved device for delivering a precise, calibrated dose of Superficial Radiation Therapy (SRT) to treat keloids caused by surgery or injury. This prospective study has been designed to focus on recurrence rates and associated treatment variables of the SRT-100™ for the treatment of recurrent keloid scars.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of keloid(s)
* Independently scheduled for treatment with SRT-100™, SRT-Vision™ or SRT-100+™ for one or more keloids
* Subject voluntary provides written consent to be in the study

Exclusion Criteria:

* Lesions of etiology other than keloids
* Any factor(s) that in the professional opinion of the investigator warrants the individual unsuitable for study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises males and females of any age who are voluntarily scheduled to be treated with the SRT-100™, SRT-Vision™ or SRT-100+™ for one or more recurrent keloids.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-08-16 (Estimated); Study Completion 2020-08-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of keloid recurrence rates. | 2 years
  Recurrence rate are calculated as the percentage of keloids that recurred at the treatment site following treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: William I Roth, MD, Principal Investigator
Locations (1):
- Dermatology and Dermatological Surgery, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No